CLINICAL TRIAL: NCT03368274
Title: To Evaluate the Clinical Efficacy of Iguratimod in the Treatment of IgG4 Related Disease (IgG4-RD) With Mild Symptom
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wen Zhang (Other)
Responsible Party: Sponsor-Investigator, Wen Zhang, professor, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IgG4-RD Iguratimod
Record Dates: First submitted 2017-09-20; First posted 2017-12-11 (Actual); Last update posted 2018-04-11 (Actual); Status verified 2018-04

CONDITIONS: IgG4-related Disease
MeSH Terms: conditions — Immunoglobulin G4-Related Disease | interventions — T 614; betamethasone dipropionate, betamethasone sodium phosphate drug combination

STUDY DESIGN:
Intervention Model Description: To compare IgG4-RD responder index, serum parameters and blood lymphocytes subpopulations at baseline and after treatment of 12 weeks and 24 weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Signal arm study (Experimental): Patients with mild symptom IgG4-RD are enrolled and inject one dosage of diprospan ,then take Iguratimod (T614), 25mg, Bid orally for three months. Firstly, we evaluate IgG4-RD responder index of patients at baseline and follow-up time.We collect the laboratory parameters and blood for lymphocytes subpopulations by flowcytometry.
  Interventions: Drug: T 614

INTERVENTIONS:
Drug: T 614 — Patients of IgG4-RD with mild symptoms are given one dose of diprospan and Iguratimod, 25mg, Bid.
  Other Names: diprospan

SUMMARY:
30 untreated IgG4 related disease (IgG4-RD) patients with mild symptom are enrolled in this study, and will be treated with one dose of diprospan,then take Iguratimod 25mg, Bid orally. Patient's peripheral blood will be collected at baseline, 12 weeks and 24 weeks of follow up. The clinical efficacy will be evaluated by the IgG4-RD responder index, serum immunoglobulin, IgG4 and IgE, cytokines, and peripheral blood T cell and B cell sub-populations will be measured at baseline and follow up.

DETAILED DESCRIPTION:
Glucocorticoid is the recognized first-line medication for IgG4-RD, but it has many side effects. In order to avoid long time glucocorticoids intake, patients with mild disease will be treated with Iguratimod combined with one dose of diprospan. 30 untreated IgG4-RD patients with mild symptom will be enrolled in this study, and be treated with one dose of diprospan,then take Iguratimod 25mg, Bid orally. 5 ml of patients' peripheral blood will be collected at baseline, 12 weeks and 24 weeks of follow up. At baseline and each follow-up, the clinical efficacy of treatment will be evaluated by IgG4-RD responder index, serum immunoglobulin, IgG4, immunoglobulin E (IgE), serum cytokines, such as interleukin 1, 6, and tumor necrosis factor, will be measured by ELISA, peripheral blood T cell sub-populations, B cell sub-populations and plasma cells will be measured by flow-cytometry.

ELIGIBILITY:
Inclusion Criteria:

* Mikulicz disease, with/without nasosinusitis or lymph node swelling.
* Without internal organs affected,
* With slow disease progression.

Exclusion Criteria:

* Vital organs related:including autoimmune pancreatitis,retroperitoneal fibrosis, sclerosing cholangitis, lung related, kidney affected, IgG4 related castleman's disease and hypophysitis，
* Combined with other connective disease,
* With tumors,
* Pregnancy or to be pregnant,
* Active infection, including hepatitis B virus, hepatitis C virus, and tuberculosis.
* Leucocytopenia, impairment of liver and kidney function,
* Allergy of Iguratimod, or cannot tolerate Iguratimod.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-06-01 (Estimated); Study Completion 2018-06-01 (Estimated)

PRIMARY OUTCOMES:
The change of IgG4-RD responder index before treatment and after treatment | 24 weeks
  Evaluate patients baseline and follow-up IgG4-RD responder index(disease activity)

SECONDARY OUTCOMES:
Changes of serum immunoglobulins subclass IgG4 levels | 24 weeks
  The IgG4 levels are tested routinely.
Patients serum cytokines | 24 weeks
  patients serum of cytokines detection by ELISA.
Peripheral blood lymphocytes sub-populations | 24 weeks
  Peripheral blood T,B sub-populations by flowcytometry
Side effects | 24 weeks
  Side effects, including laboratory tests will be recorded and tested.

CONTACTS AND LOCATIONS:
Overall Officials: Wen Zhang, Study Chair — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No